CLINICAL TRIAL: NCT06589024
Title: Remote STATE Training for Insomnia in Older Adults - Phase II
Brief Title: Remote STATE Training for Insomnia in Older Adults
Acronym: rSTATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSC-0702-22
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 36 treatment sessions, up to 5 sessions per week, ~36 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Sleep hygiene education
  Interventions: Other: Sleep Hygiene Education

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Training on computerized exercises that targets processing speed, attention and executive function for about 36 minutes per session, 5 sessions per week for a total of 36 sessions.
  Arms: Experimental Treatment
Other: Sleep Hygiene Education — Access to sleep hygiene education materials
  Arms: Active Comparator

SUMMARY:
This study called rSTATE (Remote STATE Training for Insomnia in Older Adults) is a Phase II study to definitively evaluate the efficacy of a computerized cognitive training program (rSTATE) designed to improve sleep regulation and brain health and extend functional independence in older adults with insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are 65 years of age or older. The inclusion age of ≥ 65 is in accordance with the FDA's Guideline for Industry Studies in Support of Special Populations (Geriatrics ICH-E7), which uses 65 as its cutoff for defining the geriatric population prone to insomnia.
2. Participants who have an Insomnia disorder diagnosis per DSM-V.
3. Participants who exhibit > 30 minutes sleep onset latency (SOL); and/or > 30 minutes wake after sleep onset (WASO).
4. Participants must be a US resident.
5. Participants who are fluent English speakers, per self-report, to ensure reasonable neuropsychological results on key assessments.
6. Participants must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse or a tablet.

Exclusion Criteria:

1. Participants who score ≥ 4 on the Cognitive Function Index (CFI).
2. Participants who self-report vision or hearing difficulties that would interfere with the ability to complete the study tasks.
3. Participants with past or present psychosis, schizophrenia, or bipolar disorder. Participants with other untreated psychiatric disorder, including substance abuse/dependence disorders.
4. Participants with a seizure disorder.
5. Participants with untreated obstructive sleep apnea, diagnosis of other sleep disorders not attributable to a primary sleep regulation problem (e.g., restless legs syndrome).
6. Participants with a recent hospitalization, ongoing chemotherapy or other cancer treatment.
7. Participants enrolled in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device, or behavioral treatment (CBTi) in the last 12-months that could affect the outcome of this study, or concurrent engagement in another insomnia treatment, per self-report. However, participation in standard treatments not known to affect sleep (e.g., occupational therapy) or use of prescribed medications (e.g., anti-depressants) is allowable if stable on medications for > 3 months.
8. Participants who are using computer-based cognitive training programs or have used it within a month of the consent date.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency | At 9 weeks and at 6 months

SECONDARY OUTCOMES:
Wake After Sleep Onset | At 9 weeks and at 6 months
Sleep Onset Latency | At 9 weeks and at 6 months
Total Sleep Time | At 9 weeks and at 6 months
Total Time in Bed | At 9 weeks and at 6 months
Total Wake Time | At 9 weeks and at 6 months
Sleep Quality | At 9 weeks and at 6 months
  Evaluated using the Insomnia Severity Index (ISI).
Patient Health Questionnaire - 8 questions (PHQ-8) Score | At 9 weeks and at 6 months
Generalized Anxiety Disorder Questionnaire - 7 questions (GAD-7) Score | At 9 weeks and at 6 months
Percentage of Time Spent in Stage N1 Sleep | At 9 weeks
Percentage of Time Spent in Stage N2 Sleep | At 9 weeks
Percentage of Time Spent in Stage N3 Sleep | At 9 weeks
Percentage of Time Spent in REM Sleep | At 9 weeks
REM Latency | At 9 weeks
Gradual-Onset Continuous Performance Task Score | At 9 weeks and at 6 months
  To measure task engagement
Complex Set-Shifting Score | At 9 weeks and at 6 months
  To measure task engagement

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation; Andrew Krystal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Posit Science Corporation, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No